CLINICAL TRIAL: NCT06264245
Title: Users of Remote Conferencing and Compression of Sound Dynamics : Auditory Effects
Acronym: COMPRESSED
Status: Recruiting | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut de l'Audition (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-126; 2023-A00985-40 (Other: ID RCB)
Record Dates: First submitted 2024-01-29; First posted 2024-02-16 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Auditory Perception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High exposure to compressed sound
  Interventions: Other: Audiological profile; Other: Hearing self-assessments; Other: Objective and subjective audiological tests; Other: Self-assessment of exposure sound quality
- Moderate or limited exposure to compressed sound
  Interventions: Other: Audiological profile; Other: Hearing self-assessments; Other: Objective and subjective audiological tests; Other: Self-assessment of exposure sound quality

INTERVENTIONS:
Other: Audiological profile — Video otoscopy Tympanometry High-frequency tonal audiometry
Other: Hearing self-assessments — Hearing skills questionnaire Subjective assessment of tinnitus using a visual analogue scale Self-questionnaire on the impact of tinnitus Hyperacusis self-questionnaire
Other: Objective and subjective audiological tests — Acoustic Omission Measurement of the stapedial reflex by tympanometry High-frequency tonal audiometry - exposed ear only Speech audiometry in noise Tinnitus and subjective discomfort thresholds Psychoacoustic intensity perception test
Other: Self-assessment of exposure sound quality — A self-assessment of the sound quality of the manipulated sounds heard during the exhibition will be carried out during the second follow-up visit. The elements on which the participant will be asked to make a qualitative judgement will relate to intelligibility difficulties or not; background noise (these two items in the form of a mark between 0 and 10); the clear, muffled or shrill nature of the sounds, their resonant or saturated side.

SUMMARY:
The COMPRESSED project is a descriptive, bi-centric and non-invasive study carried out by the CERIAH - IDA - Institut Pasteur and the Haute École Léonard de Vinci in Brussels on volunteer participants identified in two groups :

* be subject to high exposure to compressed sound, as defined by professional participation in events on broadcast platforms using sound signal processing systems, over the last 3 years,
* be subject to moderate or limited exposure to compressed and manipulated sound, equivalent to that of a student following certain distance learning courses. on a videoconferencing platform, alternating with other face-to-face courses, with the ability to listen during breaks, which have been taught for a maximum of 2 years.

The main objective of the COMPRESSED study is to evaluate the auditory effects of exposure to manipulated sounds (compression, filtering, equalisation, accentuation, etc.) from sound distribution platforms on the auditory system of participants who are regularly exposed to these sounds as a result of their professional activity.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Age 18 or over,
* Work with platforms using sound signal processing systems,
* Fluent in English,
* Fluent in French,
* Declare that they have no hearing loss.

For participants in the high exposure group:

- Have had a professional activity over the last three years using broadcasting platforms with sound signal processing systems,

For participants in the moderate or limited exposure group:

- Have worked between one semester and two years with platforms using sound signal processing systems.

Exclusion Criteria:

* Conductive or mixed hearing loss, i.e. where the hearing loss affects both the outer and/or middle ear and the inner ear.
* Have an asymmetric hearing loss, i.e. a difference in average hearing loss between the left and right ear of more than 20 dB,
* Have a history of otitis and/or an ENT disease that permanently affects hearing (vestibular schwannoma, Ménière's disease, sudden or fluctuating deafness, congenital hypoacusis),
* Not fluent in English
* Be under guardianship,
* Deprived of liberty by judicial or administrative decision, or subject to legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with sustained exposure to compressed sounds, as defined by professional participation in broadcast platform events using sound signal processing systems, over the last 3 years, Or Subjects with moderate or limited exposure to compressed and manipulated sound, equivalent to that of a student taking distance-learning courses on a videoconferencing platform, alternating with other face-to-face courses, with the possibility of pauses in listening, exposed for a maximum of 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Hearing assessments of participants exposed to manipulated sounds after and before exposure | 2 weeks
  Measurement of the difference between the hearing assessments of participants exposed to manipulated sounds after and before exposure

SECONDARY OUTCOMES:
Audiometric thresholds in pure tone from 125 to 8000 Hz in the subject's exposed ear before and approximately one hour after exposure, | 2 weeks
  Measurement of the difference between audiometric thresholds in pure tone from 125 to 8000 Hz in the subject's exposed ear before and approximately one hour after exposure,
Difference between the threshold of the protective reflex of the auditory pathways (middle ear muscles) measured by impedancemetry in the exposed ear when a contralateral noise is presented for a few seconds. | 2 weeks
  A contralateral noise is a low-pass filtered white noise with a cut-off at 3 kHz.
Levels of otoemissions in acoustic distortion products in the exposed ear in response to pure tone sound stimuli | 2 weeks
  Comparison of the levels of otoemissions in acoustic distortion products in the exposed ear in response to pure tone sound stimuli at 65 dB SPL around 1, 2, 3 and 4 kHz, before and approximately one hour after exposure.
Tinnitus or auditory distortion (hyperacusis) reported by participants before and after exposure. | 2 weeks
  Measurement of the difference in the perception of tinnitus or auditory distortion (hyperacusis) reported by participants before and after exposure.
Effectiveness of the protective auditory reflexes (or acoustic reflexes), obtained by impedancemetry and derived from the reading of the otoemissions for each participant. | 2 weeks
  Measurement of the difference of the effectiveness of the protective auditory reflexes (or acoustic reflexes), obtained by impedancemetry and derived from the reading of the otoemissions for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Avan, MD, Principal Investigator — CERIAH
Locations (2):
- Haute Ecole Léonard De Vinci, Brussels, Belgium
- CEntre de Recherche et d'Innovation en Audiologie Humaine, Paris, France

IPD SHARING:
Plan to Share IPD: No